CLINICAL TRIAL: NCT03642314
Title: ImPrEP Sub-study - HIV Self-Testing to Increase Combination Prevention Demand in the ImPrEP Project: an Adaptative Randomized Trial
Brief Title: HIV Self-testing in Implementation PrEP Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Oswaldo Cruz Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HIV-ST
Record Dates: First submitted 2018-08-20; First posted 2018-08-22 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: HIV Prevention
Keywords: pre exposure prophylaxis; men who have sex with men
MeSH Terms: conditions — Homosexuality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Individuals receive 5 HIV Self Test kits + vouchers to secondarily distribute to MSM/TGW from their social/sexual networks. All vouchers are uniquely identified invitations for priority access to ImPrEP sites, valid to be redeemed by a 3 month period
  Interventions: Diagnostic Test: HIV self test kit
- Control (No Intervention): Individuals receive 5 vouchers to secondarily distribute to MSM/TGW from their social/sexual networks. All vouchers are uniquely identified invitations for priority access to ImPrEP sites, valid to be redeemed by a 3 month period

INTERVENTIONS:
Diagnostic Test: HIV self test kit — HIVST receptor will be invited to priority access to PrEP sites
  Other Names: HIVST
  Arms: Intervention

SUMMARY:
This is a sub-study of an ongoing PrEP study ( HIV PrEP for men who have sex with men - MSM - and transgender women - TGW: a demonstrative project in Brazil, Peru and Mexico - ImPrEP). MSM/TGW enrolled to ImPrEP Study at the selected sites, who agree to participate in this HIV Self Test (HIVST) sub-study, will be 1:1 randomized at the third study visit either to receive 5 HIVST+voucher (intervention arm) or 5 vouchers alone (control arm) to secondarily distribute into their MSM/TGW network. All vouchers are numbered invitations for priority access to individualized HIV risk assessment and combination prevention services, including PrEP, at the ImPrEP sites. Study population comprises ImPrEP participants and their referred peers. Sample size is going to be determined at an interim analysis performed when each city has enrolled 70 participants. Trial participants will be at maximum 876 (438 intervention and 438 in the control arm) MSM and TGW included in the ImPrEP Study who received PrEP for at least 6 months in the sites from Rio de Janeiro and Lima. The study is designed as a multicenter, open, adaptative, randomized trial. The main study outcome is the voucher redemption proportion by arm.

ELIGIBILITY:
Inclusion Criteria:

* individuals who were included in the ImPrEP Study
* performed at least 3 study visits,
* accepted to participate in this sub study,
* provide informed consent form

Exclusion Criteria:

* Individuals included into ImPrEP as a result of HIVST secondary distribution

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — male
Enrollment: 876 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
voucher redemption proportion by arm | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Valdilea Veloso, PhD, Study Chair — Oswaldo Cruz Foundation

IPD SHARING:
Plan to Share IPD: No